CLINICAL TRIAL: NCT01665235
Title: The Correlation Study Between Blood Pressure Variability and the Prognosis of Ischemic Stroke With Intracranial Artery Stenosis
Brief Title: Blood Pressure Variability and the Prognosis of Ischemic Stroke With Intracranial Artery Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Shi Guowen, Principal Investigator, RenJi Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RenJiH-20120804
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Blood Pressure Variability; Intracranial Artery Stenosis
MeSH Terms: interventions — Amlodipine; Angiotensin-Converting Enzyme Inhibitors; Aspirin; Clopidogrel; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- amlodipine (Active Comparator): The amlodipine - based antihypertensive treatment group (you can add a diuretic or other )
  Interventions: Drug: Amlodipine; Drug: Aspirin or Clopidogrel; Drug: Atorvastatin
- ACEI / ARB (Experimental): ACEI / ARB -based antihypertensive treatment group ( you can add the B - blockers or other)
  Interventions: Drug: ACEI / ARB; Drug: Aspirin or Clopidogrel; Drug: Atorvastatin

INTERVENTIONS:
Drug: Amlodipine — The amlodipine - based antihypertensive treatment group (you can add a diuretic or other )
  Arms: amlodipine
Drug: ACEI / ARB — ACEI / ARB -based antihypertensive treatment group ( you can add the B - blockers or other)
  Arms: ACEI / ARB
Drug: Aspirin or Clopidogrel — aspirin 100mg / d or Clopidogrel 75mg / d (anti-platelet agents)
Drug: Atorvastatin — Atorvastatin 10 - 40mg / d ( statin therapy)

SUMMARY:
Correlation study about Blood Pressure Variability and the prognosis of ischemic stroke with intracranial artery stenosis

DETAILED DESCRIPTION:
Extracranial atherosclerotic stenosis is the main reason for the European and American white ischemic stroke and transient ischemic attack,while Atherosclerotic intracranial arterial stenosis is an important reason for Asian patients with stroke ,accounting for the 33% to 51% of a etiology ratio.The latest research suggests that varying degrees of blood pressure variability can affect the risk of stroke.This study observe the relationship between blood pressure variability and prognosis of ischemic stroke patients with intracranial arterial stenosis,with cranial magnetic resonance imaging (MRI + DWI),magnetic resonance angiography and Trans-cranial Doppler(TCD) .

ELIGIBILITY:
Inclusion Criteria:

* age : ≥ 18 years of age , ≤ 75 years old
* with intracranial artery stenosis in ischemic stroke
* the diagnosis of ischemic cerebrovascular disease are in line with the diagnostic criteria developed by the Chinese Medical Association Fourth National Cerebrovascular Disease Conference
* the patient admitted to hospital receive at least one examination like cranial MRI + DWI, MRA and TCD examination, clearly associated with intracranial arterial stenosis
* MRS score ≤ 3 points

Exclusion Criteria:

* vascular , cardiac , and unknown causes or other reasons lead to ischemic stroke
* associated with significant emotional disorders, cognitive impairment or other mental disorders can not be partners
* severe occlusion of Unilateral intracranial arteries ( over 90 % ) or bilateral stenosis more than 70%
* With extracranial artery stenosis, especially carotid and vertebral artery stenosis .
* patients with extracranial artery stenosis or patients previously done neck or intracranial artery balloon dilation , stent forming surgery or carotid endarterectomy
* Incomplete clinical data collection in patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
the incidence of stroke in a follow-up period | one year

SECONDARY OUTCOMES:
blood pressure during the compliance status in a follow-up | one year
patients with blood pressure variability in a follow-up | one year
Changes in intracranial arterial stenosis and stiffness before and after the follow-up | one year
Other vascular events ( acute ischemic heart disease or vascular death ) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Guowen Shi, MD, Principal Investigator — RenJi Hospital
Locations (1):
- RenJi Hospital, Shanghai, Shanghai Municipality, China